CLINICAL TRIAL: NCT01938092
Title: Intravaginal Diazepam for the Treatment of Pelvic Pain Among Women With Pelvic Floor Hypertonic Disorder: a Double Blind, Randomized, Placebo Controlled Trial
Brief Title: Vaginal Diazepam for the Treatment of Female Pelvic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Raymond Foster (Other)
Responsible Party: Sponsor-Investigator, Raymond Foster, Principal Investigator, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1208827
Record Dates: First submitted 2013-08-30; First posted 2013-09-10 (Estimated); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Pelvic Floor Disorders; Pelvic Pain
Keywords: High-tone pelvic floor dysfunction; Spasm; Pelvic pain; Diazepam; Female; Randomized trial
MeSH Terms: conditions — Pelvic Floor Disorders; Pelvic Pain; Spasm | interventions — Diazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diazepam (Active Comparator): Participated will be instructed to insert one 10mg tablet vaginally 1-2 times per day as needed for pain.
  Interventions: Drug: Diazepam
- Placebo (Placebo Comparator): Participated will be instructed to insert one 10mg tablet vaginally 1-2 times per day as needed for pain.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diazepam
  Other Names: Valium
  Arms: Diazepam
Drug: Placebo
  Arms: Placebo

SUMMARY:
To determine the efficacy of intravaginal diazepam for the treatment of pelvic pain associated with pelvic floor hypertonic disorder.

DETAILED DESCRIPTION:
Women who are asked to participate will already be receiving a standard conservative therapy consisting of a psyllium-based bowel regimen, heat therapy, pelvic stretching exercises, and Kegel exercises. Participants will randomly be assigned by a computer-derived random number sequence (after pregnancy is ruled out) to either the treatment group (intravaginal diazepam) or the placebo group Investigators and patients will be blinded to group assignment. The placebo or diazepam tablet will be distributed to the participant in the examining room on the day of allocation. The participant will be instructed to insert the diazepam or placebo tablet into her vagina at home. The treatment group will insert the diazepam 10 mg vaginal tablet 1-2 times daily as needed in addition to the standard conservative therapy. The placebo group will receive the standard conservative therapy, and an intravaginal tablet (visually indistinguishable from diazepam) commercially produced by the university pharmacy. After 4 weeks, patients from either group will have the option of enrolling into a standard routine program (not research) of comprehensive pelvic floor rehabilitation therapy. The Visual Analog Pain Scale, Pelvic Floor Distress Inventory-20 Questionnaire, McGill Pain Questionnaire and Global Response Assessment will be completed by the participant at the initial visit, 4 weeks, 8 weeks and 12 weeks. Participants will be given the option of choosing one or more methods for returning questionnaires: electronic mail, self-addressed home envelope, or telephone call.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old
* Primary complaint of acute or chronic pelvic pain with or without dyspareunia
* Physical exam findings consistent with levator muscle spasm
* Capable of inserting tablet in vagina without use of applicator.

Exclusion Criteria:

* Chronic narcotic use
* Non-English speaking
* Currently serving a prison sentence
* Stage III or greater vaginal prolapse
* Allergies or contraindications to benzodiazepines
* Pregnant or breastfeeding
* Currently receiving comprehensive pelvic floor rehabilitation therapy and/or vaginal valium therapy
* Unwilling or incapable of inserting tablet in vagina without applicator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond T Foster, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Missouri Center for Female Continence and Advanced Pelvic Surgery, University of Missouri Health System, Columbia, Missouri, United States

REFERENCES:
- [Derived] Holland MA, Joyce JS, Brennaman LM, Drobnis EZ, Starr JA, Foster RT Sr. Intravaginal Diazepam for the Treatment of Pelvic Floor Hypertonic Disorder: A Double-Blind, Randomized, Placebo-Controlled Trial. Female Pelvic Med Reconstr Surg. 2019 Jan/Feb;25(1):76-81. doi: 10.1097/SPV.0000000000000514. PMID 29280763

RESULTS

PARTICIPANT FLOW:
Recruitment Details: urogynecology outpatient clinic patients sequentially enrolled September 2013-August 2016. Inclusion: 18+ years of age with primary complaint of acute or chronic pelvic pain, with or without dyspareunia, and hypertonicity of the levator muscles. Exclusion: pregnant, breastfeeding, previous pelvic floor therapy, contraindication to denzodiazepines
Groups:
- Diazepam: Participated will be instructed to insert one 10mg tablet vaginally 1-2 times per day as needed for pain.
  Diazepam
- Placebo: Participated will be instructed to insert one 10mg tablet vaginally 1-2 times per day as needed for pain.
  Placebo
Period: Overall Study
Arm/Group | Diazepam | Placebo
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diazepam | Placebo | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [24 to 58] | 42 [31 to 53.5] | 42 [27 to 54.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 23 | 22 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.07 [23.79 to 30.32] | 26.99 [24.26 to 37.95] | 27.07 [24.14 to 33.52]
Gravida [Median (Inter-Quartile Range); unit: number of pregnancies] | 2 [0 to 4.5] | 2 [1 to 4] | 2 [0 to 4]
Term Pregnancies [Median (Inter-Quartile Range); unit: number of full-term pregnancies] | 2 [0 to 3] | 2 [0.25 to 3] | 2 [0 to 3]
Cesarean sections [Median (Inter-Quartile Range); unit: number of cesarean sections] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Vaginal deliveries [Median (Inter-Quartile Range); unit: number of vaginal deliveries] | 1 [0 to 3] | 1 [0 to 3] | 1 [0 to 3]
Largest baby [Median (Inter-Quartile Range); unit: gm] | 3713 [3203 to 4082] | 3487 [2821 to 4068] | 3642 [2934 to 4082]
Symptom duration [Median (Inter-Quartile Range); unit: months] | 24 [3 to 72] | 30 [12 to 120] | 24 [5 to 88]
Post void residual [Median (Inter-Quartile Range); unit: mL] | 20 [10 to 50] | 35 [11.25 to 90] | 25 [10 to 60]
Prolapse [Number; unit: participants] — Population: Prolapse data unavailable for 1 diazepam and 2 placebo participants
  participants
    number analyzed (Participants) | 24 | 22 | 46
    (all) | 4 | 4 | 8
diabetes mellitus [Count of Participants; unit: Participants] | 3 | 1 | 4
Cardiovascular disease [Count of Participants; unit: Participants] | 2 | 0 | 2
Lung disease [Count of Participants; unit: Participants] | 2 | 5 | 7
Low back pain [Count of Participants; unit: Participants] | 13 | 10 | 23
Gastrointestinal disease [Count of Participants; unit: Participants] | 8 | 11 | 19
Headache [Count of Participants; unit: Participants] | 11 | 11 | 22
Neurological disease [Count of Participants; unit: Participants] | 1 | 0 | 1
Anxiety [Count of Participants; unit: Participants] | 10 | 16 | 26
Depression [Count of Participants; unit: Participants] | 9 | 14 | 23
Bipolar disorder [Count of Participants; unit: Participants] | 2 | 3 | 5
Obsterical trauma [Count of Participants; unit: Participants] | 10 | 12 | 22
Menopausal [Count of Participants; unit: Participants] | 12 | 11 | 23
Current hormone replacement therapy [Count of Participants; unit: Participants] | 2 | 2 | 4
Vaginal estrogen use [Count of Participants; unit: Participants] | 8 | 3 | 11
Hysterectomy [Count of Participants; unit: Participants] | 9 | 8 | 17
Mesh surgery [Count of Participants; unit: Participants] | 5 | 4 | 9
Smoker [Count of Participants; unit: Participants] | 9 | 8 | 17
Heavy lifting [Count of Participants; unit: Participants] | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) for Pain
Description: Ten centimeter (100 mm) linear pain scale where patients mark their self-perceived level of pain on a paper with a 10 cm line indicating that the 0 cm position indicates no pain and the 10 cm position indicates the worst pain imaginable. The score is measured as the distance between the zero position and the patient's mark is measured in cm to the nearest mm. A higher score indicates a worse outcome.
  The change in pain score is calculated by from the value at baseline minus the value at 4 weeks. Potential range is -100 to 100, with a higher value indicating a better outcome.
Time Frame: Baseline and 4 weeks
Population: After randomization, 25 patients on diazepam treatment and 24 patients on placebo provided baseline values for visual analog score (VAS) for pain. At 4 weeks treatment, 19 patients in the diazepam group and 16 patients in the placebo group provided VAS data for pain. Data from the latter group of 35 patients were analyzed.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 19 | 16
score on a scale | 50 [20 to 75] | 39 [5 to 55]
Statistical Analysis 1: Comparison: Diazepam vs Placebo; Test type: Superiority; p = 0.62, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pelvic Floor Distress Inventory-20 (PFDI-20) Questionnaire Score at 4 Weeks.
Description: The Pelvic Floor Distress Inventory-20 is both a symptom inventory and a measure of the degree of bother and distress (quality-of-life) caused by pelvic floor symptoms. Includes 20 questions and 3 scales. Each of the 3 scales is scored from a minimum score of 0 (least distress) to a maximum of 100 (greatest distress), thus a higher score indicates a poorer outcome. The scores from each of the 3 scales are added together to give a summary score (range 0 to 300). The PFDI-20 questionnaire was administered at baseline and at 4 weeks of treatment. The outcome was the score at 4 weeks of treatment.
Time Frame: 4 weeks
Population: After randomization, 25 patients on diazepam treatment and 24 patients on placebo provided baseline values for the pelvic floor distress inventory-20 (PFDI-20) questionnaire. At 4 weeks treatment, 19 patients in the diazepam group and 16 patients in the placebo group provided PFDI-20 questionnaire data. Data from the latter group of 35 patients were analyzed.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 19 | 16
score on a scale | 96 [56 to 116] | 107 [45 to 164]
Statistical Analysis 1: Comparison: Diazepam vs Placebo; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: McGill Pain Questionnaire Score (PRI) at 4 Weeks
Description: The McGilll pain questionnaire is a validated instrument that assigns quantitative value to qualitative descriptions of chosen by the patient. The minimum pain score is 0 (would not be seen in a person with true pain) and the maximum pain score: 78. The higher the pain score the greater the pain and the poorer the outcome. measured at 4 weeks.
Time Frame: 4 weeks
Population: After randomization, 25 patients on diazepam treatment and 24 patients on placebo provided baseline values for the McGill pain questionnaire. At 4 weeks treatment, 19 patients in the diazepam group and 16 patients in the placebo group provided McGill pain questionnaire data. Data from the latter group of 35 patients were analyzed.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 25 | 24
score on a scale | 34 [28 to 38] | 33 [21 to 41]
Statistical Analysis 1: Comparison: Diazepam vs Placebo; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Diazepam | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 4/25 | 4/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diazepam (N=25) | Placebo (N=24)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
drowsiness (Nervous system disorders) | 1 (1) | 1 (1)
site irritation (Product Issues) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
1. 92% of participants Caucasian; results may differ in diverse populations
2. participants in placebo group more likely to use vaginal estrogen
3. Powered to detect a 20% difference if present; underpowered to detect a smaller difference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT01938092/Prot_SAP_000.pdf